CLINICAL TRIAL: NCT00773422
Title: The Effect of Naltrexone and Varenicline on Alcohol-Mediated Smoking Lapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sherry McKee, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: HIC0710003188; P50AA015632 (NIH)
Record Dates: First submitted 2008-10-14; First posted 2008-10-16 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Smoking
Keywords: smoking lapse behavior; smoking cessation; varenicline; naltrexone; medication effect on smoking lapse behavior
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Naltrexone; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- naltrexone + varenicline (Experimental): naltrexone (25mg) + varenicline (2mg)
  Interventions: Drug: naltrexone; Drug: varenicline
- varenicline (Experimental): varenicline 2mg
  Interventions: Drug: varenicline
- placebo (Placebo Comparator): placebo control
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: naltrexone — 25 mg/day, with 1-week lead-in medication period. The starting dose is 0 mg/day for days 1-3, followed by 12.5mg/day for day 4, followed by 25mg/day for days 5-7, plus during the laboratory session (day 8).
  Arms: naltrexone + varenicline
Drug: varenicline — 2mg/day, with 1-week lead-in medication period. The starting dose is 0.5mg/day for days 1-2, followed by 0.5mg twice daily for days 3-5, followed by 1.0 mg twice daily for days 6-7, plus during the laboratory session (day 8).
  Other Names: Chantix
  Arms: naltrexone + varenicline; varenicline
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to examine how medications thought to attenuate the effects of alcohol (naltrexone) and smoking cessation medications (varenicline) affect the ability to resist smoking and also subsequent ad-lib smoking, following a low-dose alcohol priming drink, in non-treatment seeking alcohol-drinking daily smokers.

ELIGIBILITY:
Inclusion Criteria:

* ages 21-55
* ability to read and write in English
* alcohol-drinking smokers

Exclusion Criteria:

* any significant current medical conditions that would contraindicate smoking
* current DSM-IV abuse or dependence of other substances, other than nicotine dependence or alcohol abuse.
* positive test result at intake appointments on urine drug screens conducted for opiates, cocaine, or benzodiazepines
* women who are pregnant or nursing
* suicidal, homicidal or evidence of current severe mental illness
* participants prescribed any psychotropic drug in the 30 days prior to study enrollment
* blood donation within the past 6 weeks
* individuals seeking treatment for smoking cessation or drinking or have attempted to quit smoking or drinking within the past 3 months
* specific exclusion for administration of naltrexone not specified above including chronic pain conditions necessitating opioid treatment, and evidence of significant hepatocellular injury as evidenced by SGOT or SGPT > 3x normal or elevated bilirubin
* known allergy to varenicline or taking H2blockers (e.g., Cimetidine)
* participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current protocol

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation, Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone + Varenicline | Varenicline | Placebo
Started | 11 | 9 | 10
Completed | 11 | 9 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone + Varenicline | Varenicline | Placebo | Total
Number analyzed (Participants) | 11 | 9 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.91 (8.99) | 37.67 (10.85) | 33.20 (9.73) | 33.33 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 9 | 7 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Latency to Initiate Ad-lib Smoking Session
Description: Time to smoking during the smoking delay task. Smoking delay task occurred on day 8 of the study. Range of time delay is 0 minutes to 50 minutes.
Time Frame: day 8
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Naltrexone + Varenicline | Varenicline | Placebo
Number analyzed (Participants) | 11 | 9 | 10
minutes | 28.134 (5.328) | 45.861 (6.238) | 21.737 (6.043)

2. Secondary Outcome: Number of Cigarettes Smoked During the Ad-lib Period
Description: Number of cigarettes smoked during the ad libitum phase of the smoking delay task. Task occurred on day 8 of the study.
Time Frame: day 8
Measure: Mean (Standard Error); unit: cigarettes
Arm/Group | Naltrexone + Varenicline | Varenicline | Placebo
Number analyzed (Participants) | 11 | 9 | 10
cigarettes | 1.283 (0.283) | 0.959 (0.331) | 2.23 (0.331)

ADVERSE EVENTS:
Arm/Group | Naltrexone + Varenicline | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 3/11 | 5/9 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone + Varenicline (N=11) | Varenicline (N=9) | Placebo (N=10)
Nausea/vomiting (Gastrointestinal disorders) | 2 | 2 | 1
Headache (General disorders) | 0 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1
Abnormal dreams (General disorders) | 1 | 0 | 1
Abdominal pain (General disorders) | 2 | 3 | 1
Erratic Behavior (General disorders) | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 4 | 0
Dry mouth (General disorders) | 0 | 2 | 1
Insomnia (General disorders) | 1 | 1 | 0
Difficulty Breathing (General disorders) | 0 | 1 | 1
Tight chest (General disorders) | 1 | 1 | 1
Fast heartbeat (Cardiac disorders) | 0 | 1 | 0
Suicidal Thoughts (General disorders) | 0 | 0 | 0
Depressed Mood (General disorders) | 0 | 1 | 0
Appetite change (General disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No